CLINICAL TRIAL: NCT01413022
Title: Phase IB Study of FOLFIRINOX Plus PF-04136309 in Patients With Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma
Brief Title: FOLFIRINOX Plus PF-04136309 in Patients With Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201201124; NCI-2011-01154 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-29; First posted 2011-08-09 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Flow Cytometry; Immunohistochemistry; PF-04136309

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (FOLFIRINOX chemotherapy) (Active Comparator): Patients receive FOLFIRINOX chemotherapy comprising of:
  * oxaliplatin 85 mg/m2 IV on Day 1
  * irinotecan 180 mg/m2 IV on Day 1
  * leucovorin 400 mg/m2 IV on Day 1
  * 5FU 400 mg/m2 bolus and 2400 mg/m2 CIVI over 46 hours beginning on Day 1
  Treatment is repeated every 14 days for 6 cycles.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil; Other: laboratory biomarker analysis; Other: flow cytometry; Other: immunohistochemistry staining method; Other: pharmacological study
- Group B (FOLFIRINOX and PF-04136309) (Experimental): Patients receive FOLFIRINOX chemotherapy comprising of:
  * oxaliplatin 85 mg/m2 IV on Day 1
  * irinotecan 180 mg/m2 IV on Day 1
  * leucovorin 400 mg/m2 IV on Day 1
  * 5FU 400 mg/m2 bolus and 2400 mg/m2 CIVI over 46 hours beginning on Day 1
  * PF-04136309 500 mg PO BID on days 1-14
  Treatment is repeated every 14 days for 6 cycles.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil; Other: laboratory biomarker analysis; Other: flow cytometry; Other: immunohistochemistry staining method; Other: pharmacological study; Drug: PF-04136309

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: Irinotecan
  Other Names: Campto; Camptosar; CPT-11; U-101440E
Drug: Leucovorin
  Other Names: CF; CFR; LV
Drug: Fluorouracil
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: PF-04136309
  Other Names: PF-4136309
  Arms: Group B (FOLFIRINOX and PF-04136309)

SUMMARY:
This phase I trial studies the side effects and optimal dose of PF-04136309 when given with combination chemotherapy (FOLFIRINOX; 5-fluorouracil, leucovorin, irinotecan, oxaliplatin) in treating patients with locally advanced or borderline resectable pancreatic cancer. These patients are not candidates for surgical resection which is the most effective treatment for pancreatic cancer. Giving PF-04136309 together with FOLFIRINOX may shrink pancreatic tumors in some patients so that surgery becomes an option

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To define the optimal dose and toxicity of PF-04136309 in combination with FOLFIRINOX (fluorouracil, leucovorin calcium, irinotecan hydrochloride, and oxaliplatin) in patients with borderline resectable and locally advanced pancreatic cancer.

SECONDARY OBJECTIVES:

* To evaluate the safety of PF-04136309 and FOLFIRINOX by grade 3 or 4 toxicity for clinical use.
* To determine the tumor control rate (TCR) as defined by stable disease (SD), partial response (PR), and complete response (CR): TCR = SD + PR + CR.

EXPLORATORY OBJECTIVES:

* To determine the prevalence and function of myeloid-derived suppressor cells (MDSC) in the bone marrow, peripheral circulation, and tumor before and after treatment with PF-04136309 and FOLFIRINOX.
* To determine the prevalence and function of MDSC in the bone marrow, peripheral circulation, and tumor before and after treatment with FOLFIRINOX.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed pancreatic adenocarcinoma which is borderline resectable or locally advanced; tumors considered borderline include the following: (a) no distant metastases; (b) venous involvement of the superior mesenteric vein/portal vein demonstrating tumor abutment with or without impingement and narrowing of the lumen, encasement of the superior mesenteric vein/portal vein but without encasement of the nearby arteries, or short segment venous occlusion resulting from either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection and reconstruction; (c) gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to the celiac axis; (d) tumor abutment of the superior mesenteric artery not to exceed 180 degrees of the circumference of the vessel wall
* Patient must have radiographically measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with computed tomography (CT) scan or magnetic resonance imaging (MRI) or >= 10 mm with calipers by clinical exam
* Patient myst be >= 18 years of age.
* Patient must have life expectancy of > 6 months
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count >= 1,500/mcl
  * Platelets >= 100,000/mcl
  * Hemoglobin >= 9.0 g/dL
  * Creatinine should be below the upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal limits
* Patient not on anticoagulation must have International Normalized Ratio (INR) and activated partial thromboplastin time (PTT) < 1.5 x ULN
* Patients who have had a stent placed for biliary obstruction can be included in the study
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Patient must be able to understand and willing to sign an institutional review board (IRB) approved written informed consent document

Exclusion Criteria:

* Patient must not have evidence of neuroendocrine tumor, duodenal adenocarcinoma, or ampullary adenocarcinoma
* Patient must not have a history of other malignancy =< 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix
* Patient must not have received any chemotherapy or radiation for pancreatic cancer
* Patient must not be receiving any other investigational agents
* Patient must not have brain metastases; such patients must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PF-04136309, 5FU (fluorouracil), oxaliplatin, or irinotecan
* Patient must not be on any CYP3A4 inhibitors or inducers as they may have interaction with PF-04136309 and/or irinotecan
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, any clinically active malabsorption syndrome, inflammatory bowel disease, any condition that increases the risk of severe irinotecan gastrointestinal toxicity, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not be pregnant and/or breastfeeding
* Patient must not be known to be human immunodeficiency virus (HIV)-positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Optimal dose and dose-limiting toxicity of PF-04136309 in combination with FOLFIRINOX | 28 days
  After completion of two cycles. To find the optimal dose, a 3+3 design will be used.

SECONDARY OUTCOMES:
Safety of PF-04136309 and FOLFIRINOX by grade 3 or 4 toxicity for clinical use. | 120 days (30 days after completion of treatment)
Disease response rate: TCR = SD + PR + CR | 90 days (completion of cycle 6)
Prevalence and function of MDSC in the bone marrow and tumor before and after treatment with PF-04136309 plus FOLFIRINOX or with FOLFIRINOX alone | Baseline and end of cycle 2
Prevalence and function of MDSC in peripheral circulation before and after treatment with PF-04136309 plus FOLFIRINOX or with FOLFIRINOX alone | Baseline, before cycle 2, before cycle 4, and before cycle 6

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wang-Gillam, M.D., PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Nywening TM, Wang-Gillam A, Sanford DE, Belt BA, Panni RZ, Cusworth BM, Toriola AT, Nieman RK, Worley LA, Yano M, Fowler KJ, Lockhart AC, Suresh R, Tan BR, Lim KH, Fields RC, Strasberg SM, Hawkins WG, DeNardo DG, Goedegebuure SP, Linehan DC. Targeting tumour-associated macrophages with CCR2 inhibition in combination with FOLFIRINOX in patients with borderline resectable and locally advanced pancreatic cancer: a single-centre, open-label, dose-finding, non-randomised, phase 1b trial. Lancet Oncol. 2016 May;17(5):651-62. doi: 10.1016/S1470-2045(16)00078-4. Epub 2016 Apr 4. PMID 27055731
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu